CLINICAL TRIAL: NCT02742324
Title: Phase 1/2 Randomized Trial Combination of Ruxolitinib and Peg-interferon Alpha-2a in Patients With Primary Myelofibrosis Post-polycythemia Vera-myelofibrosis or Post-essential Thrombocythemia-myelofibrosis
Brief Title: Trial Ruxolitinib and Peg-interferon Alpha-2a Combination in Patients With Primary Myelofibrosis RUXOPeg
Acronym: RUXOPeg
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUXOPeg
Record Dates: First submitted 2016-03-08; First posted 2016-04-19 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Myelofibrosis
Keywords: efficacy; safety
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolotinib and peg-IFN alpha -2a (Experimental): Phase I
  LeveL 1 Ruxolotinib 10 mg BID and peg-IFN alpha -2a 45 mcg weekly increasing doses to level 9 : Ruxolotinib 20 mg BID and peg-IFN alpha -2a 135 mcg weekly
  Phase II
  Ruxolotinib and peg-IFN alpha -2a randomized between selected doses from phase I
  Interventions: Drug: Ruxolotinib; Drug: peg-IFN alpha -2a

INTERVENTIONS:
Drug: Ruxolotinib — Ruxolitinib is administered orally twice a day (bid) everyday in 28-day treatment cycles. The starting dose is 10 mg BID and may go up to 20 mg BID. Ruxolotinib therapy starts on Cycle 1 day 1.
  Other Names: Jakavi
Drug: peg-IFN alpha -2a — Peg-IFN-alpha-2a is administered subcutaneously once a week. The doses tested are 45, 90 and 135 mcg/week. .Peg-IFN-alpha-2a therapy starts at Cycle 1Day 15.Of note, Peg-IFN-alpha-2a will only be started if the platelet count is ≥ 50x109/L at C1D15.
  Other Names: Pegasys

SUMMARY:
Phase 1/2, open-label, multi-center, trial, aiming at to identify the most efficacious dose combination that also satisfies certain safety requirements. It consists in a dose finding study to assess the safety of the combination of different doses of both ruxolitinib and peg-IFN alpha-2a, and a secondary randomized evaluation of the optimal doses found in the first part of the study to a total maximal number of 42 evaluable patients.

DETAILED DESCRIPTION:
Part 1 is a dose finding phase 1 trial that assesses the safety of the combination of different doses of both ruxolitinib and peg-IFN alpha-2a

Part 2 is a phase 2 randomized evaluation of the optimal doses found in the first part of the study to a total maximal number of 42 evaluable patients.

It will use the Bayesian Phase 1/2 adaptively randomized design proposed by Yuan and Yin (2011) for combined drugs.The trial will examine three doses of ruxolitinib: 10, 15 and 20 mg BID and three doses of the peg-IFN alpha-2a: 45, 90, and 135 mcg/week). The starting doses for each drug have been selected based on prior monotherapy experience where these doses have shown some degree of clinical activity as single agents and pharmacodynamic data supports the activity observed. In the interest of patient safety, both of these compounds will start at dose levels at or near 50% of their respective maximum tolerated doses.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Age > 18 years and < 66 years
* Diagnosis of primary or secondary myelofibrosis according to the 2008 World Health Organization (WHO) criteria for PMF (Tefferi and Vardiman 2008) and the proposed criteria for PPV-MF and PET-MF outlined by the International Working Group for Myelofibrosis Research and Treatment (Barosi et al 2008)
* Patients classified as high risk, OR intermediate risk-2, OR intermediate risk-1, as defined by the International Working Group, IWG (Cervantes, et al 2009) at diagnosis (or by the DIPSS (Passamonti et al. 2010) for patients assessed after diagnosis of PMF)
* Need for active therapy, defined as presence of at least one of the following:

  * symptomatic splenomegaly
  * presence of constitutional symptoms
  * anemia (Hb< 10g/dl)
  * leukocytosis > 25 G/l
  * thrombocytosis > 400 G/l
  * Presence of JAK2V617F , Calreticulin or MPL mutations
  * Platelet counts ≥ 150 x 109/L not reached with the aide of transfusions at screening
  * Patients with ANC ≥ 1.5 x 109/L at screening without the use of G-CSF
  * Peripheral blood blast count of ≤ 10% at Screening
  * ECOG performance status of 0, 1, or 2 at Screening
  * Negative serological Hepatitis B test (i.e. HBsAg negative and anti-HBc negative, patients positive for anti-HBc may be included if PCR for HBV DNA is negative); negative testing of Hepatitis C RNA; negative HIV test within 6 weeks prior to registration.
  * Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at Screening and effective contraception's method during the study and 75 days after the last dose.
  * Informed consent sign
  * Patients without Social Security coverage
  * Patient who is not included into another clinical study until 1 month after the end of this study

Exclusion Criteria:

* ANC < 1.5 G/l or platelets < 150 G/l
* > 10% circulating blasts
* Contra-indication to IFN alpha or to ruxolitinib
* Patients previously treated with IFN alpha or a JAK2 inhibitor
* Documented autoimmune disease at screening or in the medical history
* History or presence of depression requiring treatment with antidepressant
* Evidence of severe retinopathy (e.g. cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension)
* Thyroid dysfunction not adequately controlled
* Women of childbearing potential who have a positive serum pregnancy test at screening or who cannot or do not wish to use an effective method of contraception, during treatment and for 75 days after the last dose of study drug.
* Pregnant or nursing (lactating) women
* Patients with known active hepatitis B or C or with known HIV positivity
* Patient with a concurrent malignancy or malignancy within 3 years of Screening, with the exception of adequately treated basal or squamous cell carcinoma, non melanomatous skin cancer or curatively resected cervical cancer.
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient has active cardiac disease including any of the following:

  * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated Acquisition (MUGA) or echocardiogram (ECHO)
  * QTc> 480 msec on screening ECG (QTcF, using the Fridericia formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with documented compromise in cardiac function
  * Symptomatic pericarditis
* Patients with inadequate liver or renal function at Screening as demonstrated by:

  * encephalopathy grade 1 or more, as per West Haven Criteria
  * known hepatocellular disease (e.g. active hepatitis or cirrhosis)
  * total bilirubin> 2 x ULN and subsequent determination of direct bilirubin > 2 x ULN alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2 x ULN
* MDRD-eGFR< 45 mL/min/1.73m2 or on dialysis
* Patients who currently are willing candidates for a stem cell transplantation at the time of the screening assessments

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
study treatment efficacy/safety phase I | day 45
  Phase 1 tolerance criterion : Occurrence of dose limiting toxicities DLT within the first 45 days
study treatment efficacy/safety phase II | month 6
  Phase II Efficacy criterion: Occurrence of at least 50% reduction in spleen length as measured by palpation within the first 6 months after randomization

SECONDARY OUTCOMES:
molecular response | 12 months
  molecular response measured by the evolution of JAK2V617F or CALR or MPL mutant allele burden during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jean Jacques KILADJIAN, MD PD, Principal Investigator — FIM/GOELAMS
Locations (1):
- FILO French Innovative Leukemia Organization, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
e crf

REFERENCES:
- See also: FILO internet site — http://www.filo-leucemie.org